CLINICAL TRIAL: NCT01630317
Title: Slow Continuous Ultrafiltration Using Central vs Peripheral Line: Feasibility of Implementation, Safety and Efficacy in Acute Heart Failure Syndromes.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Nuria Ribas, Nuria Ribas, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ULISES
Record Dates: First submitted 2012-06-21; First posted 2012-06-28 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Catheterization, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peripheral acces (Experimental)
  Interventions: Procedure: Peripheral line
- Central access (Placebo Comparator)
  Interventions: Procedure: Central line vein

INTERVENTIONS:
Procedure: Peripheral line — Ultrafiltration therapy though peripheral line, two peripheral venous catheter will be placed in the arms.
  Arms: Peripheral acces
Procedure: Central line vein — Ultrafiltration therapy through central line, a central venous catheter will be placed in internal jugular or femoral vein.
  Arms: Central access

SUMMARY:
Slow continuous ultrafiltration using central vs peripheral line: feasibility of implementation, safety and efficacy in acute heart failure syndromes.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Patients hospitalized with primary diagnosis of acute heart failure defined as ≥ 2 of the following criteria:
* Peripheral or sacral edema
* Jugular venous distension or venous central pressure > 10 mmHg
* Hepatomegaly or ascites
* Pulmonary edema or pleural effusion on x-ray or pulmonary wedge pressure or end-diastolic pressure > 20 mmHg.
* High pro-BNP
* Randomization during first 24 hours
* Serum creatinine levels < 3mg/dL, and K < 6 mmol/L
* The patient should be able to communicate with research staff and meet with study procedures.
* The patient will signed informed consent.

Exclusion Criteria:

* Diagnosis of severe aortic stenosis or severe obstruction to the LVOT, tamponade, cardiac hypertrophic or restrictive cardiomyopathy.
* Impossibility of venous catheterization
* Acute coronary syndrome
* Creatinine greater than 3.0 or K greater than 6 mmol/L.
* Systolic blood pressure less than or equal to 100 mmHg
* Hematocrit greater than 45%
* Prior administration of IV vasoactive drugs in the emergency room (ER)
* Clinical instability requiring pressors during hospitalization
* Sepsis
* On or requires renal dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-11; Primary Completion 2013-10 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 48 hours after initiation of scuf therapy
  Compare patient global improvement 48 hours after initiation of scuf therapy in a group of patients with the same features treated by peripheral access against a group of patients with the same features treated by central access. This outcome will be measured by patient global assessment

SECONDARY OUTCOMES:
Security | 5th day of the study
  Compare complications in acute heart failure patients treated with scuf, in a group treated by peripheral line vs central line. This outcome will be assessed by a safety score at the AE at the 5th day of the study. ( 0 : no AE and 79 understood as the worse punctuation for the AE). Every AE has a punctuation related to the seriousness.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology Service, Hospital del Mar. Passeig Maritim 25-29,, Barcelona, Barcelona, Spain